CLINICAL TRIAL: NCT04674176
Title: The Potential Weight Loss Benefits of Rifaximin in an Intermittent Fasting Diet
Brief Title: Weight Loss Benefits of Rifaximin in an Intermittent Fasting Diet
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayhealth Medical Center (Other)
Responsible Party: Principal Investigator, Bhavin Dave, MD, Bayhealth Gastroenterology Specialist, Bayhealth Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 19901
Record Dates: First submitted 2020-10-22; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifaxamin (R) (Experimental): Patients in the experimental group will receive additional instructions to take 550 mg of Rifaximin 3 times a day for 12 days at the start of the diet. The experimental group will be provided the required doses of Rifaximin at the initial weigh-in and office visit.
  Interventions: Drug: Rifaximin
- Control (No Intervention): Participants in the control group will undergo no intervention and will only be asked to follow an Intermittent fasting diet.

INTERVENTIONS:
Drug: Rifaximin — 550 mg of Rifaximin 3 times a day for 12 days at the start of the diet.
  Arms: Rifaxamin (R)

SUMMARY:
The epidemic of overweight and obese patients presents a major challenge in chronic disease prevention and overall health across the world. Since the beginning of this century, it is considered the third most important hazard attributable to burden of disease with approximately 350 million obese people (BMI ≥30.0) and over 1 billion overweight people (BMI ≥ 25) in the world. Mechanistic studies have indicated that the microbiota influences energy utilization from the diet and influences host genes that regulate energy expenditure and storage. Thus, it is proposed that alterations in gut microbiota may play a significant role in weight loss potential.

This study seeks to expand on this idea by evaluating whether the incorporation of Rifaximin in an intermittent fasting (IF) diet plays a significant role in weight loss. Rifaximin is a nonsystemic antibiotic that works primarily in the gut to inhibit bacterial growth. It portrays unique eubiotic properties that induces a positive modulation of gut microbiota, favoring the growth of bacteria beneficial to the host without altering overall composition. Thus we propose an agent such as rifaximin would be essential in developing a positively altered gut microbiome.

Based on studies evaluating Rifaximin's role in positive gut modification, we propose that this can play a critical role in weight loss. Rifaximin may be associated with weight loss as it exerts effects that increases the concentration of bacteria more prominent in lean individuals. The choice of incorporating an intermittent fasting (IF) diet, stems from its success in prior studies. By incorporating periods of voluntary abstinence from food and drink, an IF diet has shown short term weight loss among overweight and obese people. We propose that an IF diet with an antibiotic, like Rifaximin, will create more positive alteration in gut microbiota that creates a greater potential for weight loss overall.

A group of subjects with BMI's ranging from 30-35 will be randomly selected and assigned to an experimental and control group. Each subject will be given clear instructions on how to follow a 14:10 intermittent fasting diet, in which they will fast for 14 hours and be able to eat for 10 hours a day. Patients in the experiment group will additionally receive a short-term low dosage of Rifaximin at the start of their diet. Patients will be evaluated with weekly weigh-ins and basic blood work performed at the start and at the completion of the study. The current hypothesis does not incorporate microbiome evaluation due to cost of the kits and limited funding available for the study.

DETAILED DESCRIPTION:
The epidemic of overweight and obese patients presents a major challenge in chronic disease prevention and overall health across the world. Since the beginning of this century, it is considered the third most important hazard attributable to burden of disease with approximately 350 million obese people (BMI ≥30.0) and over 1 billion overweight people (BMI ≥ 25) in the world (Mehrabani, 2018). Although there is a myriad of reasons for obesity, numerous studies have proposed that the intestinal microbiome plays an intrinsic role in overall health and obesity risk. Mechanistic studies have indicated that the microbiota influences energy utilization from the diet and influences host genes that regulate energy expenditure and storage (Davis, 2016). Thus, it is proposed that alterations in gut microbiota may play a significant role in weight loss potential.

This study seeks to expand on this idea by evaluating whether the incorporation of Rifaximin in an intermittent fasting (IF) diet plays a significant role in weight loss. Rifaximin is a nonsystemic antibiotic that works primarily in the gut to inhibit bacterial growth. It portrays unique eubiotic properties that induces a positive modulation of gut microbiota, favoring the growth of bacteria beneficial to the host without altering overall composition (Ponziani et al.,2017). In addition to its bactericidal and bacteriostatic effects, rifaximin downregulates the inflammatory response triggered by the gut microbes through inhibition of nuclear factor (NF)-kB via the pregnane X receptor (PXR) and reduces the expression of pro-inflammatory cytokines IL-1B and tumor necrosis factor alpha. These characteristics are unique to rifaximin in comparison to other antibiotics, prebiotics and probiotics (such as yogurt). These effects of rifaximin play a crucial role in gut modulation by altering bacterial virulence through inhibition of adhesion, internalization and translocation to modify bacterial metabolism (Ponziani et al.,2017). Probiotic agents such as yogurt function to increase bacterial groups (such as Bacteriodes Lactobacilli and Bifdobacteria) and there is no proven effect on gut modulation specifically. Thus we propose an agent such as rifaximin would be essential in developing a positively altered gut microbiome.

One meta-analysis investigating the associated symptoms of Rifaxamin when treating hepatic encephalopathy found weight loss to be one its side effects. (Eltawil et al.,2012). It is currently unknown whether the potential weight loss is a beneficial result of the drug or secondary to its side effects. However, based on studies evaluating Rifaximin's role in positive gut modification, we propose that this can play a critical role in weight loss. The human body is a host to vast number of microbes intrinsically linked with overall health, including obesity risk. Studies investigating the relationship between obesity and microbiota found that a low fecal bacterial diversity is associated with more marked overall adiposity, dyslipidemia, and impaired glucose homeostasis with higher low-grade inflammation. Additionally, the intestines are dominated by two divisions of bacteria: Bacteriodes and Firmictus. Within the study, obese individuals had more Firmicutes bacteria and nearly 90% less Bacteriodes than the lean individuals (Davis, 2016). This supports the reason in which Rifaximin may be associated with weight loss as it exerts effects that increases the concentration of Bifidobacteria and Bacteriodes species (Ponziani et al.,2017). By altering inflammatory cytokines, Rifaximin also plays a crucial role in improving glucose homeostasis and gut inflammation. Finally, one study investigating weight loss capabilities of rifaximin found that patients had lost a mean of 4.5 lbs in the rifaximin group compared to the control loss of 0.7lbs over a 4 month follow up (Vizuete, 2012).

The choice of incorporating an intermittent fasting (IF) diet, stems from its success in prior studies. By incorporating periods of voluntary abstinence from food and drink, an IF diet has shown short term weight loss among overweight and obese people (Ganesan et al,2018). Currently, there are no specific studies evaluating the effects rifaximin has in an IF diet. However, a meta-analysis investigating fasting diets found an alteration of gut microbiota that induced a white adipose tissue to brown adipose tissue transition - which is a beneficial reaction (Li et al, 2020). Additionally, one study investigating microbiome changes specific to a fasting diet found that there was a significantly increased abundance of Bacteriodes fragilis and Akkermansia muciniphila species (Ozkul et al, 2019). As there are already studies investigating the impact of rifaximin and fasting diet effects individually on weight loss, we propose that an IF diet with an antibiotic, like Rifaximin, will create more positive alteration in gut microbiota that creates a greater potential for weight loss overall. Although rifaximin does have some associated side effects, it is important to note that among numerous studies using Rifaximin, patients who had experienced nausea/anorexia claimed it was mild and did not withdraw from the studies (Ying et al., 2020 and Furnari 2019). Overall, this study aims to objectively determine if the use of Rifaximin with an intermittent fasting diet will improve overall weight loss results.

A group of subjects with BMI's ranging from 30-35 will be randomly selected and assigned to an experimental and control group. Each subject will be given clear instructions on how to follow a 14:10 intermittent fasting diet, in which they will fast for 14 hours and be able to eat for 10 hours a day. Patients in the experiment group will additionally receive a short-term low dosage of Rifaximin at the start of their diet. Patients will be evaluated with weekly weigh-ins and basic blood work performed at the start and at the completion of the study. It is important to note, that although we have proposed a change in gut microflora the study will focus on evaluating weight loss results and will later be followed up with another study that evaluates changes in gut microflora through microbiome testing kits. The current hypothesis does not incorporate microbiome evaluation due to cost of the kits and limited funding available for the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30-35

Exclusion Criteria:

* Underlying conditions such as hypertension, hyperlipidemia, diabetes, etc.
* BMI out of range listed above
* Inability to participate in an intermittent fasting diet
* Pregnant patients, as rifaximin should be used with caution in pregnancy due to limited data. (Subjects of childbearing age will undergo a baseline pregnancy test prior to starting the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Change from Baseline weight at 6 months
  Patients will be asked to come in for weekly weigh-ins on the same day of the week and time of day (morning, noon or evening). Weight loss will be evaluated as pounds lost or % pounds lost.
BMI | Change from Baseline BMI at 6 months
  BMI will be calculated at the beginning and at the end of the diet. Weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
HbA1C | Change from Baseline HbA1C at 6 months
  HbA1C will be measured at the start and end of the diet to evaluate percent change.
Lipids | Change from Baseline lipid results at 6 months
  Lipid panels will be evaluated at the start and end of the diet.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavin Dave, MD, Principal Investigator — Bayhealth Medical Center
Locations (1):
- Bayhealth Medical Center- Dover Family Physicians and GI Consultants Office, Dover, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis CD. The Gut Microbiome and Its Role in Obesity. Nutr Today. 2016 Jul-Aug;51(4):167-174. doi: 10.1097/NT.0000000000000167. PMID 27795585
- [Background] Eltawil KM, Laryea M, Peltekian K, Molinari M. Rifaximin vs. conventional oral therapy for hepatic encephalopathy: a meta-analysis. World J Gastroenterol. 2012 Feb 28;18(8):767-77. doi: 10.3748/wjg.v18.i8.767. PMID 22371636
- [Background] Furnari M, De Alessandri A, Cresta F, Haupt M, Bassi M, Calvi A, Haupt R, Bodini G, Ahmed I, Bagnasco F, Giannini EG, Casciaro R. The role of small intestinal bacterial overgrowth in cystic fibrosis: a randomized case-controlled clinical trial with rifaximin. J Gastroenterol. 2019 Mar;54(3):261-270. doi: 10.1007/s00535-018-1509-4. Epub 2018 Sep 19. PMID 30232597
- [Background] Ganesan K, Habboush Y, Sultan S. Intermittent Fasting: The Choice for a Healthier Lifestyle. Cureus. 2018 Jul 9;10(7):e2947. doi: 10.7759/cureus.2947. PMID 30202677
- [Background] Li L, Su Y, Li F, Wang Y, Ma Z, Li Z, Su J. The effects of daily fasting hours on shaping gut microbiota in mice. BMC Microbiol. 2020 Mar 24;20(1):65. doi: 10.1186/s12866-020-01754-2. PMID 32209070
- [Background] Mehrabani J, Ganjifar ZK (2018). Overweight and obesity: a brief challenge on prevalence, complications and physical activity among men and women.MOJ Womens Health;7(1):19-24. DOI: 10.15406/mojwh.2018.07.0016
- [Background] Ozkul C, Yalinay M, Karakan T. Islamic fasting leads to an increased abundance of Akkermansia muciniphila and Bacteroides fragilis group: A preliminary study on intermittent fasting. Turk J Gastroenterol. 2019 Dec;30(12):1030-1035. doi: 10.5152/tjg.2019.19185. PMID 31854308
- [Background] Ponziani FR, Zocco MA, D'Aversa F, Pompili M, Gasbarrini A. Eubiotic properties of rifaximin: Disruption of the traditional concepts in gut microbiota modulation. World J Gastroenterol. 2017 Jul 7;23(25):4491-4499. doi: 10.3748/wjg.v23.i25.4491. PMID 28740337
- [Background] Li Y, Hong G, Yang M, Li G, Jin Y, Xiong H, Qian W, Hou X. Fecal bacteria can predict the efficacy of rifaximin in patients with diarrhea-predominant irritable bowel syndrome. Pharmacol Res. 2020 Sep;159:104936. doi: 10.1016/j.phrs.2020.104936. Epub 2020 May 26. PMID 32470562
- [Background] Vizuete, John MD, MPH2; Randall, Charles MD1; Taboada, Carlo MD, et al (2012). Rifaximin for the Treatment of Weight Loss. American Journal of Gastroenterology, 590, Vol. 107
- [Background] Zullo A, Ridola L, Hassan C. Rifaximin therapy and Clostridium difficile infection: a note of caution. J Clin Gastroenterol. 2013 Sep;47(8):737. doi: 10.1097/MCG.0b013e31828bea4b. No abstract available. PMID 23507769